CLINICAL TRIAL: NCT04825756
Title: Evaluating the Impact of Reining in Anxiety on Childhood Anxiety
Brief Title: Evaluating the Impact of Reining in Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-00055
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Anxiety; Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): A total of up to 80 child/caregiver dyads will be enrolled in the study, anticipating that 40 dyads will complete the 10 week intervention. An equine assisted therapy called Reining in Anxiety for children with anxiety and their caregivers.
  Interventions: Behavioral: Manualized equine assisted therapy

INTERVENTIONS:
Behavioral: Manualized equine assisted therapy — This equine assisted therapy (EAT), which is delivered in a group setting, combines therapeutic horseback riding with cognitive behavioral strategies for anxiety. Each 45 minute session is delivered in a group format with up to four children between 6 and 17 years of age. Each session follows the same structure: (1) weekly review; (2) groom and connect; (3) warm-up period; (4) session activity; (5) cool down; (6) parent/caregiver psychoeducation, during which the instructor facilitates psychoeducation; and (7) homework instruction.

SUMMARY:
The purpose of this pilot study is to evaluate the impact of Reining in Anxiety for children with anxiety and their caregivers. A total of up to 80 child/caregiver dyads will be enrolled in the study, anticipating that 40 dyads will complete the 10 week intervention. The intervention will be delivered at Fieldstone Farm Therapeutic Riding Center, which is one of the largest therapeutic riding centers in the US.

DETAILED DESCRIPTION:
Reining in Anxiety is a manualized equine assisted therapy (EAT) for childhood anxiety. The manual and associated materials are being tested in this pilot study, and, if found to be successful, will be available for public consumption. This EAT, which is delivered in a group setting, combines therapeutic horseback riding with cognitive behavioral strategies for anxiety. The group meets weekly over the course of ten weeks, with each session lasting 45 minutes. Each session is delivered in a group format with up to four children between 6 and 17 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver/child dyads where the children are between six and 17 years of age and their caregivers will be enrolled in the study.
* Children must have a score of 3 or higher as measured by the GAD-2,
* Children must have a minimum level of functioning as measured by the CGAS of 41 or higher.

Exclusion Criteria:

* An inability to provide informed consent

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in levels of Anxiety | Before Session 1 (baseline) , After Session 10 ( after 6 months)
  This will be measured by the Generalized Anxiety Disorder-2 (GAD-2) questionnaire which consists of two items that assesses the presence of anxiety. Items are summed, and a score of 3 or higher is usually indicative of further evaluation.
Change in the Psychological functioning | Before Session 1 (baseline) , After Session 10 ( after 6 months)
  The Children's Global Assessment Scale (CGAS). The child is given a single score between 1- 100, based on an assessment of a range of aspects related to the child's psychological and social functioning. The score places them in one of ten categories, ranging from "extremely impaired" (1-10) to "doing very well (91-100).

SECONDARY OUTCOMES:
Change in children's emotional regulation | Before Session 1 (baseline) , After Session 10 ( after 6 months)
  This will be measured by the Children's Sadness Management Scale (CSMS) which was developed to assess children's inhibition, dysregulated expression, and coping with sadness experience and expression developed to assess three dimensions of sadness management. Children respond to 12 items on a 3-point scale (1: hardly ever, 2: sometimes, 3: often). This scale was modified to focus on dealing with anxiety rather than sadness.
Change in parents' perception of children's emotional regulation | Before Session 1 (baseline) , After Session 10 ( after 6 months)
  This is measured by the Emotion Regulation Checklist (ERC- full scale). The ERC is a 24-item questionnaire using a 4-point Likert scale that was used to assess parents' perceptions of their child's ability to manage emotion. This measure yields two empirically derived scales: (a) Emotion Regulation that assesses situationally appropriate affective displays and emotional self-awareness and (b) Lability/Negativity, which measures mood lability and culturally inappropriate affective displays. two additional questions were added about how long it takes children to regulate.
Change in emotional self efficacy | Before Session 1 (baseline) , After Session 10 ( after 6 months)
  This is measured by the Self-Efficacy Questionnaire for Children, emotional self-efficacy subscale (SEQ-C). The scale was modified the SEQ-C, which has 24 questions regarding 3 domains of self-efficacy, to utilize only the eight emotional self-efficacy items to assess parent's beliefs regarding their children's competence in controlling negative emotions. Items are scored using a 5- point Likert scale ranging from "not at all (1)" to "very well (5)." Higher scores indicate greater self-efficacy. Parents/caregivers of youth enrolled in the study completed this measure both pre and post-intervention.
Change in the level of knowledge of anxiety | Before Session 1 (baseline) , After Session 10 ( after 6 months)
  Knowledge of anxiety scale was developed by the study's researchers to assess the knowledge of anxiety from child and parent before and after the intervention, attempting to measure what has been learned in psychoeducation about anxiety.
Traumatic events of children | Before Session 1 (baseline)
  Traumatic events will be measured by the CYW Adverse Childhood Experiences Questionnaire (ACE-Q) Child, to be completed by parent/caregiver. The measure involves a list of statements of traumatic events in two sections, and parents adding up the number of statements that apply to their child. Section 1 has 10 statements, and Section 2 has 7 statements.
Perception of child's feelings to the horse | After sessions 1 (baseline), 4 (2 months), 7 (4 months), and 10 (after 6 months)
  Modified Center for the Study of Animal Wellness Scale will be used to gauge how the children feel about the horse. Attachment to the horse will be measured by the modified Center for the Study of Animal Wellness CSAW Pet B, which is a 27-item self-report measure of children's attachment. The measure presents three descriptions of feelings/perceptions about the child's relationship to the horse.
Perception of caregivers satisfaction | After Session 10 (after 6 months)
  Caregiver Satisfaction Questionnaire delivered at posttest will assess the caregiver's satisfaction with they and their child's involvement in the program
Perception of instructor's satisfaction | After Session 10 (after 6 months)
  A Satisfaction Questionnaire administered at posttest will assess the instructors' satisfaction with training and delivery of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Hoagwood, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pilot study data only

DOCUMENTS (1):
  • Informed Consent Form (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04825756/ICF_000.pdf